CLINICAL TRIAL: NCT07205315
Title: A Clinical Study Evaluating the Safety and Efficacy of GT801 Injection in Adult Patients With Relapsed/Refractory CD19-positive B-cell Hematologic Malignancies and Autoimmune Hemolytic Anemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Grit Biotechnology (Industry)
Collaborators: Zhengzhou Yihe Hospital (Unknown); Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRIT-CD-CHN-801-001
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: B-cell Acute Lymphoblastic Leukemia (B-ALL); Chronic Lymphocytic Leukemia (CLL); B-cell Non-Hodgkin's Lymphoma (B-NHL); Autoimmune Hemolytic Anemia (AIHA)
MeSH Terms: conditions — Burkitt Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell; Anemia, Hemolytic, Autoimmune

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GT801 Injection treatment group (Experimental): GT801 Injection
  Interventions: Biological: GT801 Injection

INTERVENTIONS:
Biological: GT801 Injection — GT801 Injection

SUMMARY:
The goal of this clinical study is to evaluate the safety and efficacy of GT801 injection in adult patients with relapsed/refractory CD19-positive B-cell hematologic malignancies and autoimmune hemolytic anemia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 75 years (inclusive), male or female;
* Participants with refractory or relapsed acute B-cell lymphoblastic leukemia (B-ALL), Chronic Lymphocytic Leukemia (CLL), B-cell Non-Hodgkin's Lymphoma (B-NHL) confirmed by the WHO 2016 Classification, or Autoimmune Hemolytic Anemia (AIHA) diagnosed in accordance with international consensus;
* Disease progression or recurrence after at least second-line drug treatment;
* CD19 positivity confirmed by flow cytometry and/or histopathology (excluding autoimmune hemolytic anemia);
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-1(excluding autoimmune hemolytic anemia);
* Expected survival period > 12 weeks
* For participants with hematological malignancies, the following requirements must be met:

For any prior systemic therapy (excluding immune checkpoint inhibitors), an interval of at least 2 weeks or 5 half-lives (whichever is shorter) must have elapsed between the last dose of such therapy and the planned initiation of study treatment.

For any prior treatment with immune checkpoint inhibitors (e.g., anti-PD-1/PD-L1 monoclonal antibodies such as pembrolizumab, OX40 agonists, 4-1BB agonists, etc.), an interval of at least 3 half-lives or 28 days (whichever is shorter) must have elapsed between the last dose of such treatment and the planned initiation of study treatment.

• For participants with autoimmune hemolytic anemia (AIHA), the following requirements must be met: The total course of glucocorticoid therapy shall be no less than 3 months (except for those who are unable to tolerate due to severe infection, fracture, etc.); Rituximab (100 mg or 375 mg/m²) shall be administered for at least 4 times, with hemoglobin (HB) remaining below 100 g/L at 12 weeks after the first dose; or rituximab (1000 mg per administration) shall be administered for at least 2 times, with hemoglobin (HB) remaining below 100 g/L at 12 weeks after the first dose; oral administration of any one of the following drugs including mycophenolate mofetil, cyclosporine, azathioprine, cyclophosphamide, etc., shall last for at least 4 months or be discontinued due to intolerance; intravenous therapy with fludarabine or cyclophosphamide injection shall be administered for at least 2 cycles; subcutaneous injection of bortezomib shall be administered for at least 4 times.

Exclusion Criteria:

* Participants with a history of central nervous system leukemia/lymphoma, or those with central nervous system (CNS) leukemia/lymphoma shown by magnetic resonance imaging (MRI) or PET-CT intracranial imaging during the screening period, or those with detectable malignant cells in cerebrospinal fluid or brain metastases;
* Subjects with myelofibrosis, myelodysplastic syndromes, aplastic anemia, or other malignant hematological diseases;
* Subjects with a history of or current comorbidities that cause coagulation disorders and high bleeding risk, such as disseminated intravascular coagulation (DIC), decompensated cirrhosis, esophagogastric varices, etc.;
* Subjects who experienced severe bleeding (defined as bleeding uncontrollable by medication or local therapy) within 4 weeks prior to screening, or have life-threatening bleeding (associated with thrombocytopenia) currently, or are expected to require emergency treatment within one week after enrollment;
* Subjects with secondary AIHA induced by drugs or infections;
* Subjects with hereditary hemolytic diseases or other acquired hemolytic diseases.
* Participants who undergo hematopoietic stem cell transplantation with therapeutic intent within 12 weeks of planned GT801 infusion;
* If the participant has a history of hematopoietic stem cell transplantation, the time since the participant received allogeneic hematopoietic stem cell transplantation is ≤ 6 months;
* Administration of hormonal drugs in any form within 14 days prior to infusion (except for AIHA participants requiring such drugs for hemolysis control and those receiving them for preconditioning).
* Active hepatitis B and/or active hepatitis C (HCV RNA positive); participants who are positive for hepatitis B surface antigen and/or core antibody but have HBV-DNA test results within the normal range can be included; participants who are positive for hepatitis C virus (HCV) antibody but with HCV RNA test results within the normal range are eligible for inclusion.
* Presence of central nervous system diseases or a history thereof, such as epileptic seizures, cerebrovascular ischemia/hemorrhage, dementia, cerebellar diseases, or any autoimmune diseases involving the central nervous system;
* Presence of any of the following conditions within 6 months before signing the informed consent form: uncontrolled congestive heart failure (New York Heart Association Class III-IV), angina pectoris, myocardial infarction, cardiomyopathy, stroke (except lacunar infarction), coronary/peripheral artery bypass surgery, arrhythmias with significant clinical significance (as judged by the investigator) including but not limited to ventricular arrhythmias, significantly prolonged QT interval (recommended QTc ≥ 500ms corrected by Bazett's method, specifically judged by the investigator), poorly controlled hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg), poorly controlled diabetes, pulmonary embolism, diffuse pulmonary lesions, pulmonary insufficiency, or medical conditions that the investigator deems unsuitable for the participant to participate in this clinical study;
* Prior receipt of gene-modified or gene-edited cellular therapy products (except for autologous immune cell therapy products without gene modification or editing, provided that the interval from the last administration to the first dose of GT801 is more than 1 year).
* A history of autoimmune diseases (such as Crohn's disease, rheumatoid arthritis, systemic lupus) that caused end-organ damage or required systemic immunosuppression/systemic disease-modifying agents within the past 2 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants experiencing dose limiting toxicity | 28 days
  Proportion of participants experiencing dose limiting toxicity (DLT) within 28 days after cell infusion
Incidence and severity of adverse events | From infusion to the end of the treatment at 12 months
  Incidence and severity of adverse events per NCI-CTCAE version 5.0

SECONDARY OUTCOMES:
3rd month Overall response rate (ORR) of hematological malignancy | From the date of infusion to the 3rd month
  The proportion of all evaluable subjects who were determined by the investigators to have achieved confirmed partial remission or complete remission at the third month after treatment initiation
Best Overall Response (BOR) of hematological malignancy | Up to 12 months post infusion
  Best Overall Response (BOR) refers to the best therapeutic effect recorded from the start of treatment until disease progression or recurrence.
Duration of Response (DoR) of hematological malignancy | Up to 12 months post infusion
  To evaluate the duration from the date that criteria are met for complete response or partial response as assessed by the investigator until the date of disease progression or death due to any cause
Progression-free survival (PFS) of hematological malignancy | Up to 12 months post infusion
  To evaluate the time from the date of infusion to the date of disease progression as assessed by the investigator or the date of death due to any cause
Overall survival (OS) of hematological malignancy | From the date of infusion to date of death due to any cause, or up to 12 months post infusion (whichever occurs first)
  To evaluate the time from the date of infusion to the date of death due to any cause
Overall response rate (ORR) of Autoimmune Hemolytic Anemia (AIHA) | Up to 12 months post infusion
  To evaluate the percentage of participants who have a confirmed partial response or complete response among total number of evaluable participants as assessed by the investigator
Complete Response Rate (CRR) of Autoimmune Hemolytic Anemia (AIHA) | Up to 12 months post infusion
  Complete Remission Rate (CRR) refers to the proportion of evaluable subjects who achieve complete remission following post-treatment assessment.
Partial Response Rate (PRR) of Autoimmune Hemolytic Anemia (AIHA) | Up to 12 months post infusion
  Partial Remission Rate (PRR) refers to the proportion of evaluable subjects who achieve partial remission following post-treatment assessment.
Disease-Free Recurrence (DFR) of Autoimmune Hemolytic Anemia (AIHA) | Up to 12 months post infusion
  DFR refers to the state where complete remission of the disease is achieved after treatment, all relevant medications are successfully discontinued, and stable disease without recurrence is maintained for a certain period.
Time to Response (TTR) of Autoimmune Hemolytic Anemia (AIHA) | Up to 12 months post infusion
  TTR refers to the interval from the start of treatment to the first documentation of a participant achieving a predefined response.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Zhengzhou Yihe Hospital, Zhengzhou, Henan
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No